CLINICAL TRIAL: NCT05747222
Title: Evaluation of the Effectiveness of Action Observation Theraphy (AOT) in Patients with Severe Acquired Brain Injury (sABI).
Brief Title: Action Observation Theraphy in Severe Acquired Brain Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PADUA LUCA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4599
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-12

CONDITIONS: Acquired Brain Injury
Keywords: Acquired Brain Injury; Disorder of Consciousness; Action Observation Therapy
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Action Observation Therapy (G-AOT) (Experimental): G-AOT patients will carry out AOT therapy in addition to conventional rehabilitation therapies. In case of bilateral clinical engagement, treatment with AOT will have been conducted on the limb that on motor outcome measures appears less involved.
  G-AOT patients will undergo rehabilitation treatment with AOT once a day, 5 days a week. 15 sessions will then be given, for a total duration of 3 weeks of experimental treatment with AOT.
  Interventions: Other: Action Observation Tharapy; Other: Conventional Therapy
- Group Conventional (G-CONV) (Active Comparator): G-CONV patients will only carry out rehabilitation treatments as per clinical practice.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Action Observation Tharapy — Using a 13-inch tablet, the patient will be shown, from a third-person lateral perspective framing the palmar side of the hand, a video that repeatedly plays a simple movement of daily life (grasping a glass on the table with the hand and bringing it closer to oneself) for 5 consecutive minutes. The video should be customized based on the side being treated (ex: right hemiparesis, video framing a right hand). After 1 minute of rest, the therapist will ask the patient to perform the newly observed movement for a minimum duration of 2 minutes and a maximum of 5 minutes. The cycle will be repeated a total of 3 times, for total treatment time between 25 and 35 minutes per session.
  Arms: Group Action Observation Therapy (G-AOT)
Other: Conventional Therapy — Conventional treatment will focus on joint mobilization, muscle stretching, and neuromuscular facilitation activities, using the main rehabilitation methods (e.g., neurocognitive theory, Bobath Concept, Progressive Neuromuscular Facilitation, etc.).

SUMMARY:
Action Observation Therapy (AOT) is a rehabilitation technique, used for several years, aimed at the recovery of motor function in patients with neurological and orthopedic conditions.

The essential element of this approach is the patient's observation and subsequent mime of a sequence of daily actions, aimed at achieving a goal. This task is proposed repeatedly during a single rehabilitation session and repeated for a set number of sessions. The recovery of the presented motor patterns has, as its ultimate goal, the improvement of autonomy in activities of daily living (ADLs).

The neurophysiological mechanism underlying motor cortical recovery is related to the activation of mirror neuron circuits and includes mechanisms of neuronal plasticity. In fact, it is well known how motor brain areas injured by a pathological process are able to activate during tasks of imagining or observing movements, with a correspondence between the type of movement observed and the specific motor cortical region involved in the given action. Activation of the brain areas in charge of movement, in addition to keeping the uninjured networks functioning, stimulates the injured ones by promoting, by mechanisms of neuronal plasticity, a reorganization of the primary motor cortex. The physiological basis for motor learning would thus be established, the cortical reorganization being decisive for the formation of a motor memory of the observed gesture and allowing the reacquisition, even partial, of the function of the injured motor cortex. Finally, motor cortical stimulation has a function in preventing dysfunctional cortical reorganization that intervenes after inactivity or disuse. As revealed by systematic review studies on the subject, the protocols used are very heterogeneous in terms of the type of patients to whom they were offered, the type and number of actions shown during treatments, their duration, and the rating scales used.

DETAILED DESCRIPTION:
However, in the context of patients with neurological diseases, studies have mainly been conducted on patients with outcomes of stroke, infant cerebral palsy, and Parkinson's disease. Very few data are available in the literature on the possible efficacy of AOT in patients with severe acquired brain injury (sABI).

The advantage of AOT is that it represents a method that is noninvasive, requires readily available and low-cost instrumentation, is undemanding in terms of time and resources, and for whose application there are no known adverse reactions.

In light of the above, the purpose of the study is to evaluate the application and effectiveness of rehabilitative treatment with AOT in patients with sABI of different etiology.

The research hypotheses consist of: (i) improvement of motor function assessed by clinical and functional scales (ii) improvement of cerebral cortical activation, particularly in terms of improvement of basic rhythmic frequencies and connectivity, assessed by EEG method, after rehabilitative treatment with AOT in patients with outcomes of sABI.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years;
* Having presented with a documented coma state with Glasgow Coma Scale (GCS) values ≤ 8, for at least 24 consecutive hours;
* Minimal Consciousness State (MCS) or emergence from Minimal Consciousness State (eMCS)
* Presence of muscle activity in at least one upper limb,
* Traumatic, cerebrovascular, anoxic, infectious, metabolic etiology;
* Time since acute event: 1 - 4 months;
* Unilateral or bilateral clinical involvement;

Exclusion Criteria:

* Patients in a comatose or vegetative state (VS)
* premorbid history of psychiatric or neurological conditions;
* concomitant presence of sepsis, coma, or other medical conditions that severely alter the patient's health status;
* Changes in therapy, during the study period, that may affect vigilance status (antiepileptic drugs, antidepressants, etc.) or spasticity;
* Presence of upper limb fractures;
* Level of spasticity Ashworth modified≥ 3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Motricity Index Upper Limb (MI-UL) | Change from baseline MI-UL at 3 weeks
  MI-UL can be used to assess the motor impairment in a patient who has had a stroke.
  Test for each upper limb:
  1. pincer grip
  2. elbow flexion
  3. shoulder abduction
  For the pincer grip:
  0 points, no movement 19 points, grip possible but not against gravity 33 points, normal grip
  For all other items:
  0 points, no movement 14 points, Visible movement but not for the entire joint range or against gravity 19 points, movement possible for the entire joint range against gravity but not against resistance 33 points movement performed with normal force Each segment has a total score obtained by adding the value "1" to the score of each individual item. The total score then ranges from 1 (no movement) to 100 (normal movement).

SECONDARY OUTCOMES:
Motor Assessment Scale (MAS) | Change from baseline MAS at 3 weeks
  MAS is a performance-based scale used to assess the level of impairment and daily motor function in stroke patients. It consists of 9 items to assess areas of motor function. Each item, with the exception of the item on "general tone," is assessed with a 7-point scale (0 to 6, where 6 indicates optimal motor behavior).
  For the general tone item, scoring is based on continuous observations during the assessment. A score of 4 on this item indicates a consistently normal response, a score > 4 indicates persistent hypertone, and a score < 4 indicates varying degrees of hypotone.
  Item scores (except for general tone) are summed to obtain an overall score (out of 48 points).
  For MAS 1 to 5, completion of a higher-level item suggests success in the lower-level items, and thus the lower items can be skipped.
  The upper limb section (MAS 6-8) should be scored non-hierarchically, i.e., each item within the subsets should be scored regardless of its position in the hierarchy.
Nine Hole Peg Test (9HPT) | Change from baseline 9HPT at 3 weeks
  9HPT is used to measure finger dexterity in patients with different neurological diagnoses. The patient should take the 9 pegs from a container, one by one, and to insert them into the holes in the board, as quickly as possible, using only the hand to be evaluated. After that, the patient should remove the pegs from the holes, one at a time, and reinsert them into the container.
  The evaluator should start the stopwatch as soon as the patient touches the first peg. The evaluator should stop the stopwatch when the last peg is in the container.
Coma Recovery Scale-revised (CRS-r) | Change from baseline CRS-r at 3 weeks
  CRS-r is an assessment tool that examines 6 functions: auditory, visual, oral-verbal motor, communicative, and vigilance.
  Its different items are organized hierarchically (low scores represent reflex activities, high scores describe cognitively mediated behaviors).
  For each function examined, the diagnosis of Vegetative State, Minimal Consciousness State, Emergence from Minimal Consciousness State can be made.
Level of Cognitive Functioning (LCF) | Change from baseline LCF at 3 weeks
  LCF is a tool that assesses the level of cognitive and behavioural recovery. It consists of 7 items ranging from 1=no response to 8=final-appropriate.
Glasgow Outcome Scale-Extended (GOS-E) | Change from baseline GOS-E at 3 weeks
  The Glasgow Outcome Scale- Extended (GOS-E) ranks global outcomes in TBI survivors.
  The GOS-E consists of a series of discrete categories arranged in a hierarchy and does not involve the summation of individual item scores. Choice items in the hierarchy are used to decide an outcome.
  The 8 categories are: Dead, Vegetative State, Lower Severe Disability, Upper Severe Disability, Lower Moderate Disability, Upper Moderate Disability, Lower Good Recovery, and Upper Good Recovery.
Disability Rating Scale (DRS) | Change from baseline DRS at 3 weeks
  DRS is an assessment tool for level of consciousness and functional recovery. It consists of four domains:
  (i) Vigilance, awareness and responsiveness (0 to 12 points) (ii) Cognitive ability for self-care activities (0 to 9 points) (iii) Functional level (0 to 5 points) (iv) employability (0 to 3 points). A higher score corresponds to greater disability. The overall score ranges from 0 to 30 and allows the identification of 10 categories ranging from category 1 (no disability) to category 10 (death).
Pittsburgh Partecipation Rating Scale (PPRS) | Change from baseline PPRS at 3 weeks
  The PRPS is a 6-point Likert-type measure of observed patient participation in a therapy session. The PRPS, with a full description of each anchor point, is as follows:
  Poor: The patient refused or did not participate in at least half of the session.
  Fair: The patient did not complete most of the exercises. Good: The patient participated in all exercises with good effort and completed most but not all of the exercises, and passively followed directions.
  Very good: the patient participated in all exercises with maximum effort and finished all exercises.
  Excellent: the patient participated in all exercises with maximum effort, completed all exercises and took an active interest in the exercises and/or future therapy sessions.
Electrocortical Activity | Change from baseline EEG at 3 weeks
  The information inherent in the assessment of electrocortical activity, using the electroencephalogram (EEG), asking the patient to move the treated limb (or, if not possible, to imagine the movement). The presence of a cortical potential in motor area will be assessed by following the somatotopic organization, by reconstructing a brain map in amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Luca Padua, MD, phD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy